CLINICAL TRIAL: NCT06224179
Title: Ultrasound Guided Oblique Subcostal Transversus Abdominis Plane Block(TAP) Versus Both Subcostal and Posterior TAP Block as Postoperative Analgesia in Hepatectomy
Brief Title: Role of Ultrasound Guided Transversus Abdominis Plane Block in Pain Control After Hepatectomy
Acronym: U/STAP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Ahmed wagih Ezzat deusouky, lecturer of anesthesia, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: M S 96/2021
Record Dates: First submitted 2024-01-17; First posted 2024-01-25 (Actual); Last update posted 2024-01-30 (Actual); Status verified 2024-01

CONDITIONS: Analgesia
MeSH Terms: conditions — Agnosia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group A (Experimental): Group A received ultrasound guided subcostal TAP block with 30 ml of local anesthetics and additives
  Interventions: Procedure: ultrasound guided subcostal TAP block
- Group B (Experimental): Group B received ultrasound guided both subcostal and posterior TAP block with 30 ml of local anesthetics and additives at each side
  Interventions: Procedure: ultrasound guided combined posterior and subcostal TAP block

INTERVENTIONS:
Procedure: ultrasound guided subcostal TAP block — patients will be randomly divided into two groups using a computer generated random number chart.
  Group A received ultrasound guided subcostal TAP block,
  Arms: Group A
Procedure: ultrasound guided combined posterior and subcostal TAP block — patients will be randomly divided into two groups using a computer generated random number chart.
  Group B received ultrasound guided combined posterior and subcostal TAP block,
  Arms: Group B

SUMMARY:
Inadequately managed acute pain following abdominal surgery originates from somatic pain signals in the abdominal wall and is linked to various unfavorable postoperative outcomes. These consequences encompass patient distress, respiratory complications, delirium, myocardial ischemia, extended hospital stays, an elevated risk of chronic pain, heightened analgesic consumption, delayed bowel function, and an increased need for rescue analgesics.

This study aims to assess the postoperative analgesic efficacy of ultrasound-guided Transversus Abdominis Plane (TAP) block using oblique subcostal and posterior approaches in hepatectomy.

DETAILED DESCRIPTION:
Pain control is vital to achieve enhanced recovery after abdominal surgeries . TAP block had been demonstrated to improve pain related outcomes after abdominal surgeries.

Postoperative pain management for patients undergoing hepatic resection is a challenge due to the risk of perioperative liver dysfunction.TAP block is a promising regional analgesic technique. This study aimed to evaluate the effect of US-guided subcostal approach versus combination of both subcostal and posterior approaches of TAP block

The patients will be randomly divided into two groups :

group A will recieve oblique subcostal TAP block and group B will recieve both subcostal and posterior TAP block .

ELIGIBILITY:
Inclusion Criteria:

* ASA I and II patients. aged 18 to 50 years. 70 to 80 kg.

Exclusion Criteria:

* patients under 18 years of age.

  * History of Allergic reactions to study drugs.
  * Opioid or analgesic abuse, and chronic treatment with opioids, or non-steroidal anti-inflammatory drugs.
  * History of bleeding tendency or coagulopathy .

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-02-01 (Estimated); Primary Completion 2024-05-01 (Estimated); Study Completion 2024-06-01 (Estimated)

PRIMARY OUTCOMES:
postoperative analgesia (VAS) during the 1st 24 hours in ICU | 24 hours
  Pain will be assessed on admission and at 2, 4, 8, 12 and 24 hours at rest and with passive flexion of hip and knee joint using visual analogue scale (VAS) ranging from 0 for no pain to 10 for worst pain.